CLINICAL TRIAL: NCT03407651
Title: Phase 2 Study to Evaluate the Pharmacokinetics, Efficacy and Safety of a Daily Subcutaneous Treatment Regimen With Marzeptacog Alfa (Activated) for Bleeding Prophylaxis in Adult Subjects With Hemophilia A and B Subjects With an Inhibitor
Brief Title: Study of Coagulation Factor VIIa Variant Marzeptacog Alfa (Activated) in Adult Subjects With Hemophilia A and B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalyst Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MAA-201
Record Dates: First submitted 2018-01-04; First posted 2018-01-23 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-06

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia B With Inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1a (Experimental): Coagulation Factor VIIa variant, 18 µg/kg by intravenous route
  Interventions: Biological: Coagulation Factor VIIa variant
- Part 1b (Experimental): Coagulation Factor VIIa variant, 30 µg/kg by subcutaneous route
  Interventions: Biological: Coagulation Factor VIIa variant
- Part 2 (Experimental): Coagulation Factor VIIa variant, 30, 60, 90, 120 µg/kg by subcutaneous route
  Interventions: Biological: Coagulation Factor VIIa variant

INTERVENTIONS:
Biological: Coagulation Factor VIIa variant — Single intravenous injection of MarzAA, followed by single subcutaneous injection of MarzAA, followed by daily subcutaneous injection of MarzAA for 50 days at final dose level required.

SUMMARY:
Phase 2, multi-center, open-label study designed to evaluate the PK, bioavailability, PD, efficacy and safety of a daily subcutaneous [SC] treatment regimen with MarzAA for bleeding prophylaxis in 12 adult subjects with hemophilia A or B with an inhibitor and history of frequent spontaneous bleeding episodes.

DETAILED DESCRIPTION:
Multi-center, open-label Phase 2 study to evaluate the PK, bioavailability, PD, efficacy and safety of a daily SC treatment regimen with MarzAA for bleeding prophylaxis in adult subjects with hemophilia A or B with an inhibitor. The study will enroll and dose, both intravenously and subcutaneously, a total of 12 adult male subjects with severe congenital hemophilia A or B with an inhibitor, and history of frequent bleeding episodes during the 6 months prior to enrollment, as per the individual's bleeding and treatment records.

Once a subject is enrolled into the trial, the study will be conducted in three parts (occurring consecutively):

Part 1a (24 hours): Single IV administration of MarzAA; Part 1b (48 hours): Single SC administration of MarzAA; Part 2: Daily SC administration. Dose escalation in Part 2 will occur if breakthrough bleeding occurs. Subjects are treated for 50 days at the final dose level required.

ELIGIBILITY:
Inclusion Criteria:

* Severe congenital hemophilia A or B with an inhibitor.
* History of frequent spontaneous bleeding episodes.
* Male, age 18 or older.
* Affirmation of informed consent with signature confirmation before any trial-related activities.

Exclusion Criteria:

* Receiving prophylaxis treatment.
* Previous participation in a clinical trial evaluating a modified rFVIIa agent.
* Known positive antibody to FVII or FVIIa detected by central laboratory at screening.
* Have a coagulation disorder other than hemophilia A or B.
* Significant contraindication to participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, MD, PhD, MMM, Study Director — Catalyst Biosciences
Locations (9):
- Hematology Center after Prof. R. Yeolyan, Yerevan, Armenia
- Georgia (3):
  - JSC "K.Eristavi National Center of Experimental and Clinical Surgery", Tbilisi
  - LTD M.Zodelava Hematology Centre, Tbilisi
  - LTD Medinvest - Institute of Hematology and Transfusiology, Tbilisi
- Gabinet Lekarski, Bartosz Korczowski, Rzeszów, Poland
- Russia (3):
  - Regional Clinical Hospital, Kemerovo
  - FGU Kirov Scientific Research, Kirov
  - Center for Hemophilia Treatment, Saint Petersburg
- Haemophilia Comprehensive Care Centre, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No
This is an open label study so each investigator will have full access to all study subject data that is entered into the database

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11 subjects participated in the study.
Groups:
- Overall Study Population: Period 1: Part 1a
  Coagulation Factor VIIa variant, 18 µg/kg by intravenous route
  Coagulation Factor VIIa variant: Single intravenous injection of MarzAA, followed by single subcutaneous injection of MarzAA, followed by daily subcutaneous injection of MarzAA for 50 days at final dose level required.
  Period 2: Part 1b
  Coagulation Factor VIIa variant, 30 µg/kg by subcutaneous route
  Coagulation Factor VIIa variant: Single intravenous injection of MarzAA, followed by single subcutaneous injection of MarzAA, followed by daily subcutaneous injection of MarzAA for 50 days at final dose level required.
  Period 3: Part 2
  Coagulation Factor VIIa variant, 30, 60, 90, 120 µg/kg by subcutaneous route
  Coagulation Factor VIIa variant: Single intravenous injection of MarzAA, followed by single subcutaneous injection of MarzAA, followed by daily subcutaneous injection of MarzAA for 50 days at final dose level required.
Period: Period 1: Part 1a
Arm/Group | Overall Study Population
Started | 11
Completed | 10
Not Completed | 1
Period: Period 2: Part 1b
Arm/Group | Overall Study Population
Started (One subject completed Part 1a of the study and opted to enter into Part 2 of the study and did not enter Part 1b, making the number of subjects in Part 1b smaller than the number of subjects in Part 1a. That subject withdrew consent after 1 SC dose in Part 2 but is counted as a discontinuation in Part 1 as no additional assessments were performed and the subject did not enter Part 1b. One subject had poor IV access and skipped Part 1b of the study.) | 9
Completed | 9
Not Completed | 0
Period: Period 3: Part 2
Arm/Group | Overall Study Population
Started | 11 (The subject who discontinued after 44 daily SC doses in Part 2 elected to participate in Period 3.)
Completed | 8
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: Safety Population
Arm/Group | Safety Population
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] — This assessment was not available for one subject in the study. Population: Safety Population
  cm
    number analyzed (Participants) | 10
    (all) | 171.57 (11.061)
Weight [Mean (Standard Deviation); unit: kg] — This assessment was not available for one subject in the study. Population: Safety Population
  kg
    number analyzed (Participants) | 10
    (all) | 69.05 (21.255)
BMI [Mean (Standard Deviation); unit: kg/m^2] — This assessment was not available for one subject in the study. Population: Safety Population
  kg/m^2
    number analyzed (Participants) | 10
    (all) | 23.091 (5.1478)

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Episode Prevention Success
Description: Annualized bleed rate (ABR; spontaneous and total) during Part 2 when on final MarzAA dose level versus recorded historical ABR. The analysis of the primary endpoint (annualized bleeding rate ABR for spontaneous and traumatic bleeds) of the final dose of MarzAA each subject was treated was based on the 1-sample test compared to a predefined rate assumed for the on-demand therapy. The latter was assumed to be 12 (or 1 bleed per month), which was the minimum ABR for each subject according to inclusion criterion 2 (defined as the H0), with no maximum value. A higher score indicated a worse outcome. ABR is on a scale of 0 to 365, with a lower score reflective of a lower number of bleeding events in a year.
Time Frame: Day 1 of final MarzAA dose level - Day 50
Population: Overall number of participants analyzed was based on the Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part 2: MarzAA 30 and 60 µg/kg by subcutaneous route
  Single intravenous injection of MarzAA, followed by single subcutaneous injection of MarzAA, followed by daily subcutaneous injection of MarzAA for 50 days at final dose level required.
Arm/Group | Part 2
Number analyzed (Participants) | 10
score on a scale | 1.4640 (3.08638)

2. Secondary Outcome: Occurrence of Breakthrough Bleeding
Description: Occurrence of breakthrough bleeds requiring escalation to higher dose level
Time Frame: From Day 5 of dose level until occurrence of event
Population: Single intravenous injection of MarzAA, followed by single subcutaneous injection of MarzAA, followed by daily subcutaneous injection of MarzAA for 50 days at final dose level required. Overall number of participants analyzed was based on the Intent-to-Treat Population.
Measure: Number; unit: number of breakthrough bleeds
Groups:
- Part 1a, MarzAA IV 18 µg/kg: Single intravenous injection of MarzAA 18 µg/kg
- Part 1b, MarzAA SC 30 µg/kg: Single subcutaneous injection of MarzAA 30 µg/kg
- Part 2, MarzAA 30 µg/kg: MarzAA 30 µg/kg by subcutaneous injection daily for 50 days
- Part 2, MarzAA 60 µg/kg: MarzAA 60 µg/kg by subcutaneous injection daily if dose escalation required, up to Day 50
Arm/Group | Part 1a, MarzAA IV 18 µg/kg | Part 1b, MarzAA SC 30 µg/kg | Part 2, MarzAA 30 µg/kg | Part 2, MarzAA 60 µg/kg
Number analyzed (Participants) | 10 | 9 | 11 | 2
number of breakthrough bleeds | 0 | 0 | 5 | 0

3. Secondary Outcome: Occurrence of Clinical Thrombotic Event
Description: Occurrence of clinical thrombotic event not attributable to another cause
Time Frame: From date of first dose until date of first occurrence of clinical event, assessed up to treatment Day 50
Population: as for outcome 2
Measure: Number; unit: number of events
Groups:
- Part 1, MarzAA IV 18 µg/kg: Single intravenous infusion of MarzAA 18 µg/kg
- Part 1, MarzAA SC 30 µg/kg: Single subcutaneous infusion of MarzAA 30 µg/kg
Arm/Group | Part 1, MarzAA IV 18 µg/kg | Part 1, MarzAA SC 30 µg/kg | Part 2, MarzAA 30 µg/kg | Part 2, MarzAA 60 µg/kg
Number analyzed (Participants) | 10 | 9 | 11 | 2
number of events | 0 | 0 | 0 | 0

4. Secondary Outcome: Coagulation Assessment - Prothrombin Time
Description: Change in coagulation parameter (prothrombin time [PT]) from pre-dose. Min-max values are reflective of the highest and lowest values for all measured timepoints.
Time Frame: From date of pre-dose to 24 hours (Part 1a), pre-dose to 48 hours (Part 1b), and pre-dose to Day 50 (Part 2)
Population: as for outcome 2
Measure: Median (Full Range); unit: seconds
Groups:
- Part 1a, MarzAA IV 18 µg/kg: Single intravenous infusion of MarzAA 18 µg/kg
- Part 1b, MarzAA SC 30 µg/kg: Single subcutaneous infusion of MarzAA 30 µg/kg
Arm/Group | Part 1a, MarzAA IV 18 µg/kg | Part 1b, MarzAA SC 30 µg/kg | Part 2, MarzAA 30 µg/kg | Part 2, MarzAA 60 µg/kg
Number analyzed (Participants) | 10 | 9 | 10 | 2
seconds | -3.70 [-5.30 to 1.50] | -2.80 [-4.8 to -0.3] | -3.0 [-6.5 to 1.2] | -4.80 [-4.8 to 3.8]

5. Secondary Outcome: Coagulation Assessment - Activated Partial Thromboplastin Time
Description: Change in coagulation parameter (activated partial thromboplastin time [aPTT]) from pre-dose. Min-max values are reflective of the highest and lowest values for all measured timepoints.
Time Frame: From date of pre-dose to 24 hours (Part 1a), 48 hours (Part 1b), to Day 50/end of study (Part 2)
Population: as for outcome 2
Measure: Median (Full Range); unit: seconds
Arm/Group | Part 1a, MarzAA IV 18 µg/kg | Part 1b, MarzAA SC 30 µg/kg | Part 2, MarzAA 30 µg/kg | Part 2, MarzAA 60 µg/kg
Number analyzed (Participants) | 9 | 9 | 10 | 2
seconds | -10.60 [-57.4 to 140.8] | 1.30 [-30.65 to 50.1] | -8.30 [-47.3 to 30.3] | -15.00 [-20.15 to 2.0]

6. Secondary Outcome: Coagulation Assessment - Fibrinogen
Description: Change in coagulation parameter (fibrinogen) from pre-dose. Min-max values are reflective of the highest and lowest values for all measured timepoints.
Time Frame: From date of pre-dose to 24 hours (Part 1a), 48 hours (Part 1b), or Day 50 (Part 2).
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/dL
Groups:
- Part 1a: MarzAA 18 µg/kg by intravenous injection
- Part 1b: MarzAA 30 µg/kg by subcutaneous injection
- Part 2, MarzAA 60 ug/kg: MarzAA 60 µg/kg by subcutaneous injection daily if dose escalation required, up to Day 50
Arm/Group | Part 1a | Part 1b | Part 2, MarzAA 30 µg/kg | Part 2, MarzAA 60 ug/kg
Number analyzed (Participants) | 9 | 9 | 10 | 2
mg/dL | -10.0 [-173 to 51] | -15.00 [-133 to 108] | -4.0 [-112 to 146] | -4.0 [-84.0 to 116]

7. Secondary Outcome: Number of Events of Antibody Formation
Description: Occurrence of antibody formation resulting in a decreased endogenous level of coagulation Factor VII (FVII) or Factor VII activated (FVIIa)
Time Frame: From time of first dose of MarzAA until date of first occurrence of clinical event, assessed up to treatment Day 50
Population: as for outcome 2
Measure: Number; unit: number of events of antibody formation
Arm/Group | Part 1a | Part 1b | Part 2, MarzAA 30 µg/kg | Part 2, MarzAA 60 µg/kg
Number analyzed (Participants) | 10 | 9 | 11 | 2
number of events of antibody formation | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Events of an Antibody Response
Description: Occurrence of an antibody response to MarzAA and whether it is inhibitory and cross-reactive to wild-type recombinant coagulation FVII (wt-rFVII) or wt-FVIIa.
Time Frame: From time of first dose of MarzAA until date of first occurrence of clinical event, assessed up to treatment Day 50.
Population: as for outcome 2
Measure: Number; unit: number of events of antibody response
Arm/Group | Part 1a | Part 1b | Part 2, MarzAA 30 µg/kg | Part 2, MarzAA 60 µg/kg
Number analyzed (Participants) | 10 | 9 | 11 | 2
number of events of antibody response | 0 | 0 | 0 | 0

9. Secondary Outcome: Thrombogenicity Assessment
Description: Number of participants with clinically significant levels of thrombogenicity markers (D-dimer, Prothrombin fragment 1+2 (F1+2), and thrombin-antithrombin complex [TAT]), based on standard laboratory tests and clinical examination with a specific search for any signs of thrombosis
Time Frame: From time of pre-dose of MarzAA at Day 1 until date of first occurrence of thrombotic event, assessed up to treatment Day 50.
Population: Overall number of participants analyzed was based on the Intent-to-Treat Population.
Measure: Number; unit: participants
Groups:
- Part 1a, MarzAA IV 18 µg/kg: MarzAA 18 ug/kg by intravenous injection
- Part 1b, MarzAA SC 30 µg/kg: MarzAA 30 ug/kg by subcutaneous injection
Arm/Group | Part 1a, MarzAA IV 18 µg/kg | Part 1b, MarzAA SC 30 µg/kg
Number analyzed (Participants) | 10 | 9
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Members of the study team recorded all reportable events with start dates occurring any time after informed consent was obtained until study completion, or discharge, for non-serious AEs and until 30 days after the last day of study participation for SAEs. The duration of the study was 52 days.
Description: Adverse events and serious adverse events are based on the Safety Population.
Groups:
- MarzAA IV 18 μg/kg: IV infusion of 18 ug/kg MarzAA, Part 1 of study
- MarzAA SC 30 μg/kg: SC infusion of MarzAA SC 30 μg/kg, Part 1 of study
- MarzAA 30 ug/kg: SC infusion of MarzAA 30 ug/kg, Part 2 of study
- MarzAA 60 ug/kg: SC infusion of MarzAA 60 ug/kg, Part 2 of study
Arm/Group | MarzAA IV 18 μg/kg | MarzAA SC 30 μg/kg | MarzAA 30 ug/kg | MarzAA 60 ug/kg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 1/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 1/10 | 0/2
Other Adverse Events (participants affected / at risk) | 1/10 | 1/9 | 8/10 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MarzAA IV 18 μg/kg (N=10) | MarzAA SC 30 μg/kg (N=9) | MarzAA 30 ug/kg (N=10) | MarzAA 60 ug/kg (N=2)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MarzAA IV 18 μg/kg (N=10) | MarzAA SC 30 μg/kg (N=9) | MarzAA 30 ug/kg (N=10) | MarzAA 60 ug/kg (N=2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (10) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A planned outcome measure (coagulation assessment via MarzAA activity levels) of the protocol was not calculated as as a satisfactory assay could not be developed. Data is not reported for two allowed dose groups in Part 2, MarzAA 90 μg and 120 μg, as no subjects were treated at these dose levels

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT03407651/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT03407651/SAP_001.pdf